CLINICAL TRIAL: NCT02245230
Title: Cardiovascular Effects of Angiotensin (1-7) in Essential Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We were not able to enroll adequate number of participants that met the inclusion/exclusion criteria, and we run out of funding.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 140958
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hypertension; Hypertension, Essential
Keywords: Hypertension; Autonomic Nervous System; Renin-Angiotensin System; Angiotensin (1-7); Ganglionic Blockers; Trimethaphan; Blood Pressure; Hemodynamics
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — angiotensin I (1-7); Trimethaphan; trimethaphan camsylate; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intact Study Day (Active Comparator): Subjects will receive saline infusion for 60 minutes followed by five ascending doses of Angiotensin (1-7) ranging from 0.5 to 20 ng/kg/min. Each dose will be maintained for 10 minutes with hemodynamic measurements and blood samples collected at the end of each dosing period.
  Interventions: Drug: Angiotensin (1-7)
- Autonomic Blockade Study Day (Experimental): Autonomic blockade will be induced by continuous intravenous infusion of trimethaphan starting at 0.5-1.0 mg/min and increasing by 1.0 mg/min every 2 to 6 minutes up to an infusion rate of 5 mg/min. Blood pressure will be restored to pre-trimethaphan levels with intravenous phenylephrine infusion at individually titrated doses, starting with 0.1 ug/kg/min. Angiotensin (1-7) will then be infused in five ascending doses ranging from 0.5 to 20 ng/kg/min. Each dose will be maintained for 10 minutes with hemodynamic measurements and blood samples collected at the end of each dosing period.
  Interventions: Drug: Angiotensin (1-7); Drug: Trimethaphan; Drug: Phenylephrine

INTERVENTIONS:
Drug: Angiotensin (1-7) — Angiotensin (1-7) is a peptide produced by the body. It will be administered as an acute intravenous infusion with doses ranging from 0.5 to 20 ng/kg/min.
  Other Names: Angiotensin-(1-7); Angiotensin I (1-7)
Drug: Trimethaphan — Trimethaphan is a Nn-nicotinic receptor antagonist that blocks sympathetic and parasympathetic transmission at the level of the autonomic ganglia. It will be administered as an acute intravenous infusion with doses ranging from 0.5 to 5.0 mg/min.
  Other Names: Trimethaphan Camsylate
  Arms: Autonomic Blockade Study Day
Drug: Phenylephrine — Phenylephrine is an alpha 1-adrenergic agonist. It will be administered as an acute intravenous infusion to restore blood pressure following trimethaphan with doses ranging from 0.1 to 0.5 ug/kg/min.
  Other Names: Phenylephrine Hydrochloride
  Arms: Autonomic Blockade Study Day

SUMMARY:
The purpose of this study is to better understand the cardiovascular effects of the vasodilatory peptide Angiotensin (1-7) in human hypertension. In this study, the investigators will test the hypothesis that systemic Angiotensin (1-7) infusion produces negligible effects with intact baroreceptors, and that the cardiovascular effects of this peptide are unmasked following elimination of baroreflex buffering.

DETAILED DESCRIPTION:
Pharmacologic approaches to increase levels or actions of the vasodilatory peptide Angiotensin (1-7) are currently in development for the treatment of hypertension based on findings from animal studies. There are limited and contradictory clinical studies, however, and it is unclear if this peptide even contributes to blood pressure regulation in humans. The purpose of this study is to learn more about the cardiovascular effects of Angiotensin (1-7) in essential hypertension, and to examine interactions of this peptide with the autonomic nervous system for blood pressure regulation. The investigators propose that the difficulties in showing Angiotensin (1-7) cardiovascular effects in previous clinical studies relates to the buffering capacity of the baroreceptor reflex to prevent changes in blood pressure. In this study, the investigators will test the hypothesis that Angiotensin (1-7) produces negligible effects with intact baroreceptors, and that the cardiovascular effects of this peptide are unmasked following elimination of baroreflex buffering. To test this hypothesis, the investigators will examine the effects of acute intravenous Angiotensin (1-7) infusion on blood pressure in subjects with essential hypertension under intact conditions and following acute autonomic withdrawal with the ganglionic blocker trimethaphan. The primary outcome will be the decrease in systolic blood pressure produced by Angiotensin (1-7) infusion, with comparisons made between intact and blocked study days. As a secondary objective, the investigators will examine for changes in systemic hemodynamics and circulating hormones in response to the Angiotensin (1-7) infusion, to determine potential mechanisms underlying any changes in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 60 years of age
* Hypertension defined by two or more properly measured seated blood pressure readings >130/85 mmHg. This will allow us to include subjects with "pre-hypertension."
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Previous allergic reaction to study medications
* Evidence of type I or type II diabetes (i.e. fasting glucose >126 mg/dl, use of anti-diabetic medications)
* Cardiovascular disease other than hypertension such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* History of serious cerebrovascular disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) > 2.0 x upper limit of normal range]
* Impaired renal function (serum creatinine >1.5 mg/dl)
* Anemia (hemoglobin <13.5 g/dl in males or <12.5 g/dl in females)
* Treatment with phosphodiesterase 5 inhibitors
* Treatment with anticoagulants
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol (i.e. clinically significant abnormalities on clinical, mental examination or laboratory testing or inability to comply with protocol)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Change from baseline in systolic blood pressure over the 50-minute infusion period
  The primary outcome will be the change in systolic blood pressure from baseline produced by the Angiotensin (1-7) infusion, with comparisons made between intact and autonomic blockade study days.

SECONDARY OUTCOMES:
Hemodynamic Measures | Change from baseline in hemodynamic measures over the 50-minute infusion period
  We will examine for changes in cardiac output, stroke volume, and systemic vascular resistance to determine hemodynamic mechanisms underlying any changes in blood pressure during Angiotensin (1-7) infusion.
Circulating Renin-Angiotensin System Components | Change from baseline in circulating renin-angiotensin system components over the 50-minute infusion period
  We will examine for changes in plasma renin activity, angiotensin II, Angiotensin (1-7), and aldosterone levels to determine renin-angiotensin system hormonal mechanisms underlying any changes in blood pressure during Angiotensin (1-7) infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No